CLINICAL TRIAL: NCT02908152
Title: The Effect of Curcumin Supplement on Metabolic Factors and Hepatic Fibrosis in Nonalcoholic Fatty Liver Patients
Brief Title: Curcumin Supplement in Nonalcoholic Fatty Liver Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 467
Record Dates: First submitted 2016-09-05; First posted 2016-09-20 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes; Nonalcoholic Fatty Liver
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- curcumin (Active Comparator): curcumin
  Interventions: Dietary Supplement: curcumin
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: curcumin — 1500 mg
  1 capsule / day for 12 weeks
  Arms: curcumin
Dietary Supplement: placebo — 1500 mg
  1 capsule / day for 12 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the effects of curcumin supplement on metabolic factors and hepatic fibrosis in nonalcoholic fatty liver patients with type 2 diabetes. Subjects will participate in 3 month, two group, randomized intervention, where one group (n=25) will take 1.5g/d curcumin and the other group (n=25) will take a placebo to compare differences in outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with type 2 diabetes based on ADA definition or who only take oral antidiabetic drug;
* CAP score >263.

Exclusion Criteria:

* Taking any kind of antibiotics two weeks before recruitment;
* History of alcohol consumption;
* pregnancy or lactation;
* Professional athletes;
* Other liver disease (viral/etc);
* High dose synthetic estrogens, methotrexate, amiodarone, steroids, chloroquine, immunosuppressive drugs;
* A history of Cardiovascular disease;
* Renal disease, Celiac disease, Cirrhosis;
* History of Upper GI surgery;
* A history of hypothyroidism or Cushing's syndrome;
* History of drug dependence;
* Body mass index (BMI) ≥35 kg/m2;
* A restrictive diet or weight change ≥ 5 kg during the 3months prior to study;
* Any change in treatment with oral hypoglycemic; anti hypertensive and antilipid agents during the study;
* Use of weight loss medications.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Hepatic steatosis | [12 weeks]
  measured by CAP score using Fibroscan

SECONDARY OUTCOMES:
Glucose | [12 weeks]
HBA1C | [12 weeks]
ALT | [12 weeks]
AST | [12 weeks]

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI, Tehran, Iran